CLINICAL TRIAL: NCT01086462
Title: A Microdose Study to Describe the Intravenous Pharmacokinetics of [14C]-GSK2239633 in Healthy Male Subjects
Brief Title: Intravenous Microdose Pharmacokinetic (PK) Study With [14C]-GSK2239633
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114041
Record Dates: First submitted 2010-02-18; First posted 2010-03-15 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: GSK2239633; RADIOLABEL; PHARMACOKINETICS; INTRAVENOUS; MICRODOSE
MeSH Terms: conditions — Asthma

ARMS (1):
- GSK2239633 (Experimental): Single dose infusion of study drug over 15 minutes
  Interventions: Drug: GSK2239633

INTERVENTIONS:
Drug: GSK2239633 — 100 ug GSK2239633 containing approximately 10kBq [14C]-GSK2239633

SUMMARY:
This study is a first administration to man microdose study to describe the pharmacokinetics of GSK2239633.

DETAILED DESCRIPTION:
The different shapes of the pharmacokinetic (PK) profiles following administration of GSK2239633 in rat and dog make it difficult to reliably predict the human PK profile. This microdose study will provide an early readout on the distribution and clearance profile of the drug in man and will be used to model potential clinical oral doses. The study will be conducted using an open-label, single dose design in one group of healthy male volunteers. Each subject will receive a single intravenous infusion of 100ug GSK2239633 (containing approximately 10kBq of [14C]-GSK2239633), administered over 15 minutes. Subjects will attend for a screening visit within 30 days prior to Day 1 and receive a single dose infusion of study drug on Day 1. Blood and urine samples will be taken over 48 hours for pharmacokinetic and total radioactivity analysis, and safety and tolerability will be monitored. Subjects will be discharged on Day 3 and a follow-up telephone call will be made 4-10 days post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects are defined as individuals who in the opinion of the Investigator are free from clinically significant cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, endocrine, neurological and psychiatric disease or malignancy as determined by medical history, physical examination, laboratory studies, and other tests (including ECG). Subjects with values outside the normal range which are deemed to be clinically relevant should always be excluded from enrollment.
* Male between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* Subject must agree to use one of the contraception methods listed in Section 8.1. of the protocol. This criterion must be followed from the time of screening until 90 days after the follow up
* Body weight >or= 50 kg and BMI within range 18.5-29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Single QTcF <450 msec; or QTcF <480 msec in subjects with Bundle Branch Block
* Lifelong non-smokers or ex-smokers of greater than 6 months and <5 pack year history. Pack years = (cigarettes per day smoked/20) x number of years smoked.
* AST, ALT, alkaline phosphatase and bilirubin <or=1.5 ULN (isolated bilirubin >1.5 x ULN acceptable if bilirubin is fractionated and direct bilirubin <35%)

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* A positive pre-study drug/alcohol screen
* A positive test for HIV antibody
* History of regular alcohol consumption within 6 months of study defined as an average weekly intake of >12 units/week for males. One unit is equivalent to 8g of alcohol; a half-pint (~250ml) of beer, 1 glass (100ml) of wine or 1 (35 ml) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (including snuff, nicotine-containing gum) within 6 months prior to screening
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to first dosing: 60 days, 5 half-lives or twice the duration of the biological effect of investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Participation in a clinical trial involving administration of 14C-labelled compounds within last 12 months
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Unwillingness or inability to follow procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* A calculated creatinine clearance (Cockroft and Gault formula) of <90 mL/min
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01-21 (Actual); Primary Completion 2010-02-22 (Actual); Study Completion 2010-02-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC0-inf, Cmax, AUC0-t, t1/2, clearance, volume of distribution) of [14C]-GSK2239633 and total drug-related material | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Cahn A, Hodgson S, Wilson R, Robertson J, Watson J, Beerahee M, Hughes SC, Young G, Graves R, Hall D, van Marle S, Solari R. Safety, tolerability, pharmacokinetics and pharmacodynamics of GSK2239633, a CC-chemokine receptor 4 antagonist, in healthy male subjects: results from an open-label and from a randomised study. BMC Pharmacol Toxicol. 2013 Feb 28;14:14. doi: 10.1186/2050-6511-14-14. PMID 23448278
- See also: Results for study 114041 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114041?search=study&search_terms=114041#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register